CLINICAL TRIAL: NCT06911177
Title: Efficacy of Yeast Mannan Supplementation on Increasing Stool Frequency in Generally Healthy Adults: A Randomized Controlled Trial
Brief Title: Yeast Mannans and Stool Frequency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB202500359
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-08

CONDITIONS: Defecation Frequency
Keywords: yeast mannan; stool frequency; transit time; microbiota
MeSH Terms: interventions — bleomycin-mannan conjugate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yeast mannan supplementation (Experimental): Yeast cell wall fraction obtained from Saccharomyces cerevisiae containing mannan-oligosaccharides and mannoproteins will be supplemented at 12 g/day.
  Interventions: Dietary Supplement: Yeast mannan
- Control supplementation (Placebo Comparator): The control supplement, containing yeast protein, yeast extract, and maltodextrin, will be provided at 12 g/day.
  Interventions: Dietary Supplement: Control (placebo)

INTERVENTIONS:
Dietary Supplement: Yeast mannan — Yeast cell wall fraction of manno-oligosaccharides and mannoproteins supplemented at 12 g/day.
  Other Names: yeast cell wall fraction
  Arms: Yeast mannan supplementation
Dietary Supplement: Control (placebo) — A supplement containing yeast protein, yeast extract, and maltodextrin, provided at 12 g/day.
  Arms: Control supplementation

SUMMARY:
Findings from an open-label pilot study of 20 adults suggested that supplementation with 15 g/day of yeast mannans was highly tolerable and demonstrated specific modulation of the microbiota and increased stool frequency in a subset of subjects reporting ≤1 stool per day at baseline. The primary aim of this randomized, double-blind, controlled trial is to determine if yeast mannan supplementation at 12 g/day will increase stool frequency in generally healthy adults reporting ≤1 stool per day. Secondary aims will determine the effect of yeast mannans on intestinal transit time, gastrointestinal symptoms, fecal microbiota composition, and urinary and fecal metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* Adults who report a stool frequency of ≤ 1 per day.
* Able to provide written informed consent in English.
* Willingness to consume 1 supplement (12 g of yeast mannans or control) daily for 28 days.
* Willingness to maintain their usual diet and physical activity patterns throughout the study and refrain from the consumption of any yeast-based foods (e.g. Marmite or Vegemite) or yeast extract supplements.
* Willing to comply with study procedures, including stool and urine colle

Exclusion Criteria:

* Stool frequency of < 3 per week
* Yeast allergy
* Vegan dietary pattern
* Self-reported kidney disease
* Elite athletes or long-distance runners
* Use of antibiotic drugs within 1 month of screening
* Current use of laxatives or antidiarrheal medications
* Use of other investigational products within 3 months of the screening
* Previously or currently being treated for intestinal diseases or conditions, including irritable bowel disease (i.e., IBS-D or IBS-mixed), Crohn's disease, ulcerative colitis, celiac disease, or gastrointestinal cancer.
* Previous gastrointestinal surgery (e.g., gastric bypass, fundoplication, bowel resection).
* Current cancer treatment.
* Currently pregnant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Defecation frequency | From enrollment to the end of treatment at 6 weeks.
  Mean daily defecation frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food Science and Human Nutrition, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided